CLINICAL TRIAL: NCT03893240
Title: A Multi-Center, Low-Interventional Study With a Retrospective Component in Participants With Late-Onset Pompe Disease
Brief Title: Neutralizing Antibody Seroprevalence Study With a Retrospective Component in Participants With Late-Onset Pompe Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spark Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SPK-GAA-100
Record Dates: First submitted 2019-03-11; First posted 2019-03-28 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Pompe Disease; Pompe Disease (Late-onset); Glycogen Storage Disease Type 2; LOPD; Lysosomal Storage Diseases; Acid Maltase Deficiency
MeSH Terms: conditions — Glycogen Storage Disease Type II; Lysosomal Storage Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with Late Onset Pompe disease (Other): This is a multi-center, low-interventional study with a retrospective component in participants with LOPD. During a single study visit, assessments including but not limited to, liver health, neutralizing antibodies to SPK-3006 capsid and GAA, anti-GAA binding antibodies, GAA activity and GAA antigen levels will be performed. Additional information will be collected to provide retrospective evaluations relating to muscle and liver inflammation and/or injury. Historic data relating to Pompe disease will be collected from medical records. The retrospective and laboratory data collected may assist in providing baseline information for a future investigational gene therapy study.
  Interventions: Diagnostic Test: Neutralizing Antibody to SPK-3006 capsid

INTERVENTIONS:
Diagnostic Test: Neutralizing Antibody to SPK-3006 capsid — Collected during a single study visit to establish the occurrence of neutralizing antibodies to SPK-3006 capsid in participants with LOPD on an enzyme replacement regimen.

SUMMARY:
The purpose of this study is to obtain information pertaining to the occurrence of antibodies to investigational SPK-3006 capsid and GAA, GAA activity and GAA antigen levels in the usual care setting of Late-Onset Pompe Disease (LOPD) participants on an enzyme replacement regimen. Additionally, a careful evaluation of laboratory and functional testing in patients with LOPD may provide information to better understand the disease features and better drive the design of a future interventional investigational gene therapy trial. An understanding of the underlying status of liver and muscle health in individuals with LOPD may also inform best surveillance during the conduct of gene therapy trials.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent and authorization to use protected health information in accordance with national and local privacy regulations
* Male or females ≥18 years of age
* Currently on ERT using regular recombinant human GAA infusions for at least 18 months prior to screening
* Documented history of clinically moderate late-onset Pompe disease.

Exclusion Criteria:

* History of HIV infection
* Requires any invasive ventilation (other than BiPAP at night) or noninvasive ventilation while awake and upright
* Previously received SPK-3006
* Previously dosed with any investigational or approved gene therapy product at any time or treated with an investigational drug within the last 12 weeks (vaccination studies are accepted)
* Any concurrent clinically significant condition that would not allow the potential participant to complete the Day 1 examinations, or other condition that, in the opinion of the Investigator and/or Sponsor, makes the subject unsuitable for participation in the study
* Unable or unwilling to comply with the schedule of visits and/or study assessments described in the clinical protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2020-10-27 (Actual)

PRIMARY OUTCOMES:
Neutralizing Antibodies Titer to SPK-3006 capsid | 1 day
  The neutralizing antibodies titer to SPK-3006 is measured once prospectively at one site visit.
Occurrence of Neutralizing Antibodies to SPK-3006 capsid | 1 day
  The proportion of participants who have Neutralizing Antibodies to SPK-3006 capsid.

SECONDARY OUTCOMES:
Anti-GAA binding antibodies Titer | 1 day
  Anti-GAA binding antibodies titer is measured once prospectively at one site visit.
Occurrence of Anti-GAA binding antibodies across participants | 1 day
  The proportion of participants who have Anti-GAA binding antibodies.
Neutralizing antibodies to circulating GAA Titer | 1 day
  Neutralizing antibodies to circulating GAA titer is measured once prospectively at one site visit and, if available, retrospectively from medical records that are within 24 months of signing the informed consent.
Occurrence of Neutralizing antibodies to circulating GAA | 1 day
  The proportion of participants who have neutralizing antibodies to circulating GAA.
GAA activity level | 1 day
  GAA activity level (percent of normal) is measured once prospectively at one site visit and, if available, retrospectively from medical records that are within 24 months of signing the informed consent.
GAA antigen level | 1 day
  GAA antigen level (percent of normal) is measured once prospectively at one site visit and, if available, retrospectively from medical records that are within 24 months of signing the informed consent.

CONTACTS AND LOCATIONS:
Overall Officials: Tahseen Mozaffar, MD, Principal Investigator — University of California Irvine Health
Locations (18):
- United States (6):
  - Barrow Neurological Institute, Phoenix, Arizona
  - University of California Irvine Health, Orange, California
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Minnesota Medical School, Minneapolis, Minnesota
  - Oregon Health & Science University, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
- France (3):
  - Hôpital Raymond-Poincaré, Garches, Hauts-de-Seine
  - Assistance Publique Hôpitaux de Marseille, Marseille
  - CHU Nice, Nice
- Klinikum der Universität München, München, Germany
- Italy (6):
  - Università degli Studi di Messina, Messina
  - Universita degli Studi di Milano - Clinica Oculistica I, Milan
  - Università degli Studi di Napoli Federico II, Napoli
  - Fondazione Mondino Istituto Neurologico Nazionale a Carattere Scientifico, Pavia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Azienda Ospedaliera Universitaria Citta della Salute e della Scienza di Torino, Torino
- Erasmus University Medical Center, Rotterdam, Netherlands
- Salford Royal NHS Foundation Trust, Salford, United Kingdom

IPD SHARING:
Plan to Share IPD: No